CLINICAL TRIAL: NCT02938559
Title: Can the Memory Support Intervention Improve Depression Outcome Following Cognitive Therapy?
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Allison Harvey, Professor of Clinical Psychology,, University of California, Berkeley
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: R01MH108657 (NIH)
Record Dates: First submitted 2016-10-06; First posted 2016-10-19 (Estimated); Last update posted 2021-02-02 (Actual); Status verified 2021-01

CONDITIONS: Depressive Disorder, Major
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Cognitive Behavioral Therapy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Cognitive Therapy plus Memory Support (Experimental)
  Interventions: Behavioral: Cognitive Therapy (CT) for depression + Memory Support
- Cognitive Therapy-as-usual (Active Comparator)
  Interventions: Behavioral: Cognitive Therapy (CT) for depression

INTERVENTIONS:
Behavioral: Cognitive Therapy (CT) for depression — There is evidence that CT for major depressive disorder (MDD) can be as effective as antidepressant medication for the initial treatment of moderate to severe MDD. Moreover, following the withdrawal of treatment, patients treated with CT are significantly less likely to relapse than patients treated with antidepressant medication and CT is at least as effective as antidepressant medication in preventing subsequent relapse. CT aims to alter the symptomatic expression of depression and reduce risk for subsequent episodes by correcting the negative beliefs and maladaptive information processing presumed to underlie the disorder and alter the systematic tendency to misperceive reality in a pessimistic fashion.
  Arms: Cognitive Therapy-as-usual
Behavioral: Cognitive Therapy (CT) for depression + Memory Support — The Memory Support Intervention will be delivered interwoven with CT. The Memory Support Intervention is designed to improve patient memory for treatment and involves a series of specific procedures that support the encoding and retrieval stages of episodic memory. It is comprised of eight memory promoting strategies: attention recruitment, categorization, evaluation, application, repetition, practice remembering, cued-based reminder and praise recall. These strategies are proactively, strategically and intensively integrated into treatment-as-usual to support encoding. Memory support is delivered alongside each 'treatment point', defined as a main idea, principle, or experience that the treatment provider wants the patient to remember or implement as part of the treatment.
  Arms: Cognitive Therapy plus Memory Support

SUMMARY:
The aim of this study protocol is to conduct a confirmatory efficacy trial to test whether the Memory Support Intervention improves illness course and functional outcomes in major depressive disorder (MDD) and cognitive therapy (CT).

DETAILED DESCRIPTION:
Background. Major depressive disorder (MDD) is one of the most prevalent psychiatric disorders and a leading cause of disability worldwide. Existing therapies fail to produce complete recovery. Progress toward improving outcome must include innovations that are safe, powerful, inexpensive and simple (for fast and effective dissemination). The proposed research seeks to test one such innovation. The investigators seek to improve outcome by improving memory for the content of cognitive therapy (CT) sessions. CT is one of the most promising approaches to the treatment of MDD, yet there is room for improvement.

It is proposed that adding memory enhancing strategies to CT may improve MDD outcome because: (a) MDD is often characterized by memory impairment, (b) there is evidence that the memory impairment is modifiable, (c) CT typically entails the activation of emotion, (d) emotion can impair or bias memory and (e) there is evidence that memory for the content of therapy sessions is poor.

Hence, the overall goal is to evaluate if integrating strategies designed to enhance memory for the content of CT sessions improves treatment outcome for MDD. Cognitive support involves a series of specific procedures that support the encoding and retrieval stages of an episodic memory. It is hypothesized that CT+Memory Support, relative to CT-as-usual, will be associated with improved illness course and functional outcome at the end of treatment as well as 6 and 12 months post-treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age 18+ years
* Willing and able to give full consent
* English language fluency
* Diagnosis of major depressive disorder (MDD), first episode, recurrent or chronic, according to DSM-5
* Minimum score 26 or above on the Inventory of Depressive Symptomatology, Self-Report (IDS-SR). This cutoff denotes at least 'moderate' depression
* If taking medications for mood, medications must be stable for the past four weeks

Exclusion Criteria:

* History of Bipolar Disorder
* History of Psychosis or psychotic features
* Lifetime history of failure to respond to 4 or more sessions of CBT/CT for depression
* Current non-psychotic disorder if it constitutes the principal diagnosis and if it requires treatment other than that offered in the project. 'Principal' is defined as the disorder currently most distressing and disabling, using a widely accepted severity rating scale capturing distress and interference (0-8, 4+ indicates clinical severity)
* Moderate or severe substance use in the past 6 months where 'moderate' is defined as 4-5 symptoms and 'severe' is defined as 6+ listed in DSM-5 for each of the substance-related disorders
* Evidence of any medical disorder or condition that could cause depression, preclude participation in CT, or is associated with memory problems, that is not currently stabilized and/or managed under the care of a physician or the presence of an active and progressive physical illness or neurological degenerative disease,
* Current suicide risk sufficient to preclude treatment on an outpatient basis (assessed by the Columbia-Suicide Severity Rating Scale) or current homicide risk (assessed by our staff, a case manager or psychiatrist)
* Pregnancy or breastfeeding
* Not able/willing to participate in and/or complete the pre-treatment assessments

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 178 (Actual)
Dates: Start 2016-11; Primary Completion 2020-08-05 (Actual); Study Completion 2020-08-05 (Actual)

PRIMARY OUTCOMES:
Remission | Post-Treatment which is two weeks after final therapy session (i.e. 18-20 weeks after initial intake interview)
  % Remission is defined as signs and symptoms must be absent or close to it for >=3 weeks and operationalized as IDS-SR less than 14.
Relapse at 6 Months | Calculated at 6-months after the end of treatment [the end of treatment is defined as two weeks after the final therapy session (i.e. 18-20 weeks after the initial intake interview
  % Relapse is defined as 'return to an MDE following remission' and operationalized as greater than or equal to 14 on the IDS-SR at follow-up for those who had remitted.
Relapse at 12 Months | Calculated at 12 months after the end of treatment [the end of treatment is defined as two weeks after the final therapy session (i.e. 18-20 weeks after the initial intake interview
  % Relapse is defined as 'return to an MDE following remission' and operationalized as greater than or equal to 14 on the IDS-SR at follow-up for those who had remitted.
Functional Impairment | Change from pre-treatment to post-treatment defined as two weeks after the final therapy session (i.e. 18-20 weeks after the initial intake interview) to 6-month follow-up to 12-month follow-up
  WHODAS 2.0 total score
Patient Memory for Treatment | Week 4, Week 8, Week 12, Week 16 of treatment as well as Post Treatment, defined as two post-treatment defined as two weeks after the final therapy session (i.e. 18-20 weeks after the initial intake interview) to 6-month follow-up to 12-month follow-up
  Cumulative Recall on the Patient Treatment Recall Task
Generalization Task | Week 4, Week 8, Week 12, and Week 16 of treatment as well as Post Treatment, defined as two weeks after the final therapy session (i.e. 18-20 weeks after the initial intake interview) to 6-month follow-up to 12-month follow-up
Declarative Memory | Change from pre-treatment to post-treatment defined as two weeks after the final therapy session (i.e. 18-20 weeks after the initial intake interview) to 6-month follow-up to 12-month follow-up
  Hit Rate minus False Alarm Rate minus Lure Rate on the Episodic Face-Name Learning Task
Working Memory | Change from pre-treatment to post-treatment defined as two weeks after the final therapy session (i.e. 18-20 weeks after the initial intake interview) to 6-month follow-up to 12-month follow-up
  No. of correct hits minus the no. of false positives on 3-Back of the N-Back
Memory Support | 20-26 sessions of treatment (over 16 weeks) spanning 18-20 weeks after initial intake interview
  Total Amount on the Memory Support Rating Scale on randomly selected therapy tapes.

SECONDARY OUTCOMES:
Response to Treatment | Post-Treatment which is two weeks after final therapy session (i.e. 18-20 weeks after initial intake interview)
  % Response is defined as a clinically significant degree of symptom reduction and operationalized as 50% reduction in pre-treatment symptom severity on the IDS-SR.
Magnitude of symptom change is operationalized as change on IDS-SR | Change from Pretreatment to Post-Treatment
Recovery | Calculated at 6-months and 12-months after the end of treatment [the end of treatment is defined as two weeks after the final therapy session (i.e. 18-20 weeks after the initial intake interview
  % Recovery is defined as 'remission sustained for >=4 months' and is operationalized via the LIFE.
Recurrence | Calculated at 6-months and 12-months after the end of treatment [the end of treatment is defined as two weeks after the final therapy session (i.e. 18-20 weeks after the initial intake interview
  % Recurrence is defined as 'return to an MDE following recovery' and is established using the SCID.
Time to relapse or recurrence | Calculated at 6-months and 12-months after the end of treatment [the end of treatment is defined as two weeks after the final therapy session (i.e. 18-20 weeks after the initial intake interview
  Time to relapse or recurrence following response or remission will be established using the SCID.
Functional Impairment | Change from pre-treatment to post-treatment defined as two weeks after the final therapy session (i.e. 18-20 weeks after the initial intake interview) to 6-month follow-up to 12-month follow-up
  4-question Healthy Days core module
Patient Memory for Treatment | Change from pre-treatment to post-treatment defined as two weeks after the final therapy session (i.e. 18-20 weeks after the initial intake interview) to 6-month follow-up to 12-month follow-up
  Past Session Recall on the Patient Treatment Recall Task
Working Memory | Change from pre-treatment to post-treatment defined as two weeks after the final therapy session (i.e. 18-20 weeks after the initial intake interview) to 6-month follow-up to 12-month follow-up
  No. of correct hits minus the no. of false positives on 0-Back, 1-Back, 2-Back of the N-Back
Memory Support | 20-26 sessions of treatment (over 16 weeks) spanning 18-20 weeks after initial intake interview
  Number of Types on the Memory Support Rating Scale
Competencies of Cognitive Therapy Scale (CCTS) (Exploratory) | Post Treatment, defined as two weeks after the final therapy session (i.e. 18-20 weeks after the initial intake interview), 6 month Follow-Up, 12 month Follow-Up
  Measure of patient competence at using cognitive therapy skills.

OTHER OUTCOMES:
Pre-Treatment Assessment Telephone Screen to determine Eligibility | Pre-Treatment
Structure Clinical Interview for DSM-5 (SCID) | Pre-Treatment as well as Post Treatment, defined as two weeks after the final therapy session (i.e. 18-20 weeks after the initial intake interview), 6 month Follow-Up, 12 month Follow-Up
Quick Inventory for Depressive Symptomatology-Self-Report (QIDS) | At the beginning of every treatment session (i.e., for 18-20 weeks after the initial intake interview)
IQ National Adult Reading Test (NART) | Pre-Treatment
Treatment Provider Recall Task | Week 4, Week 8, Week 12, Week 16, and last session of treatment, defined as 16-18 weeks after the initial intake interview
Medication (medication type and dosage) | Duration of Study which is at the pre-treatment assessment, at the post-treatment which defined as two weeks after the final therapy session (i.e., 18-20 weeks after the initial intake interview), at the 6-month follow-up and at the 12-month follow-up.
Other Treatment/Therapy Tracking Log (presence/absence) | Duration of Study which is at the pre-treatment assessment, at the post-treatment which defined as two weeks after the final therapy session (i.e., 18-20 weeks after the initial intake interview), at the 6-month follow-up and at the 12-month follow-up.
Credibility/Expectancy Questionnaire (CEQ) | Treatment Week 2 and 2 weeks Post-Treatment, at the 6-month follow-up and at the 12-month follow-up
Patient usefulness and utilization of cognitive therapy skills scale (Exploratory) | 2 weeks post-treatment, 6-post-treatment, 6-month follow-up, and 12-month follow-up
  Measure completed by patients indicating how useful they found specific cognitive therapy skills, and how often they used each skill.
Patient Conceptualization of Depression Task (Exploratory) | pre-treatment, post-treatment, 6-month follow-up
Treatment Adherence Rating Scale-Therapist Version | After each treatment session filled out by therapist (20-26 times)
Memory Support Treatment Provider Checklist | After treatment sessions in weeks 4, 8, 12, and 16 filled out by therapist (4 times)
Memory Support Rating Scale | Week 1, Week 4, Week 8, Week 12, Week 16 of treatment

CONTACTS AND LOCATIONS:
Locations (1):
- University of California, Berkeley, Berkeley, California, United States

REFERENCES:
- [Derived] Sarfan LD, Zieve G, Gumport NB, Xiong M, Harvey AG. Optimizing outcomes, mechanisms, and recall of Cognitive Therapy for depression: Dose of constructive memory support strategies. Behav Res Ther. 2023 Jul;166:104325. doi: 10.1016/j.brat.2023.104325. Epub 2023 May 13. PMID 37210887
- [Derived] Gumport NB, Zieve GG, Dong L, Harvey AG. The Development and Validation of the Memory Support Treatment Provider Checklist. Behav Ther. 2021 Jul;52(4):932-944. doi: 10.1016/j.beth.2020.11.005. Epub 2020 Dec 17. PMID 34134832